CLINICAL TRIAL: NCT02599142
Title: A Randomised Controlled Trial Comparing the Accuracy and Acceptability of Closed-face and Open-face Thermoplastic Immobilisation Shells in Cranial Radiotherapy
Brief Title: Comparing Immobilisation Shells in Cranial Radiotherapy
Acronym: CORIOLIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR4362
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Brain Metastases; Bone Metastases; Brain Tumor, Primary; Brain Tumor Adult; Brain Tumor - Metastatic
Keywords: radiotherapy immobilisation; open-face shells
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Single centre parallel group randomised controlled trial investigating the impact of using open-face thermoplastic immobilisation shells upon setup reproducibility in patients having cranial radiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Closed-face shells (Active Comparator): Cranial radiotherapy using the control closed-face immobilisation shell.
  Interventions: Device: Group A: Closed-face shell
- Group B: open-face shell (Experimental): Cranial radiotherapy using the experimental open-face immobilisation shell
  Interventions: Device: Group B: Open-face shell

INTERVENTIONS:
Device: Group A: Closed-face shell — As for arm description
  Arms: Group A: Closed-face shells
Device: Group B: Open-face shell — As for arm description
  Arms: Group B: open-face shell

SUMMARY:
Patients having radiotherapy to their head and neck wear an immobilisation shell to prevent patient movement and improve treatment accuracy. These shells tend to cover the face and have the potential to cause anxiety and distress in patients, particularly if they suffer with claustrophobia or a similar fear. The study will use an 'open-face' shell that does not cover the face and compare this with the investigators' current 'closed-face' shell. The investigators will obtain treatment verification x-ray images to assess the daily set-up errors and compare these between the two shell type, and ask both patients and radiographers of their experiences from using the shells.

Hypothesis: Open-face immobilisation shells offer equivalent accuracy and efficiency of radiotherapy delivery and are better accepted by patients and radiographers as compared to closed-face immobilisation shells for cranial radiotherapy.

DETAILED DESCRIPTION:
Patients will be randomised into one of two groups, with group A acting as the control group using the investigators' standard 3--point closed--face shell, and group B using the 3--point open--face shell (experimental group). Each procedure is discussed with the patient before commencement. Patients will be positioned into the optimal treatment position and the shell will be fabricated as per manufacturer instructions by pre-treatment radiographers. This is followed by the patient having a planning CT scan of their head while wearing their shell to allows radiographers and doctors to localise and plan the treatment. At the end of this appointment, the patient will be asked to complete the first of three questionnaires regarding their experience of wearing the shell. Radiographers will be asked to complete a questionnaire of their experience of using the shell, and complete timing data for the procedures.

On the first day of treatment, radiographers will discuss the treatment process and side effects of treatment with the patient, and treatment will be delivered under current department protocols using linear accelerators (linacs). During the course of the treatment, radiographers will obtain 5 sets of verification images for the study, and these will be assessed for set-up errors as per current department policy. Where possible, treatment fields will be used to verify patient position to keep radiation doses from verification imaging as low as reasonably practicable (ALARP). Patients will be asked to complete two more questionnaires on their experience, one on their first day and one on their last day of treatment. Radiographers will also complete questionnaires on these days. Timing data will be obtained for all treatment fractions.

The patient's perspective of the planning and treatment processes will be almost identical to that of patients having cranial radiotherapy that are not in the trial. The only differences that will be observed will be the use of an open-face shell (for patients in group B), completion of three questionnaires, and additional verification imaging.

ELIGIBILITY:
Inclusion Criteria:

* patients prescribed cranial radiotherapy using virtually simulated parallel opposed fields with:
* 5 or more fractions of virtually simulated cranial radiotherapy
* treatment for Primary Central Nervous System Lymphoma (PCNSL), prophylactic cranial irradiation (PCI), or primary or secondary cerebral or bony lesions

Exclusion Criteria:

* patients unable to give informed consent
* patients requiring conformal or inverse-planned radiotherapy
* patients requiring stereotactic radiotherapy
* patients who have previously had cranial or head and neck radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Assessment of treatment verification imaging to determine inter-fraction reproducability of immobilisation shells | within 2 weeks of completion of treatment
  Assessment of verification imaging to determine individual systematic and random errors. Individual errors are collated to determine group systematic and random errors for comparison.

SECONDARY OUTCOMES:
Timing data | within 2 weeks of patient completion of treatment
  Completion of data on time taken for setup, imaging, and total appointment time
Assessment of imaging to determine intra-fraction motion | within 2 weeks of patient completion of treatment
  Comparison of verification imaging with in-treatment imaging records to determine magnitude of intra-fraction motion. These will be assessed per patient and compared between both groups.
Patient acceptance and tolerability of immobilisation shells (pre-treatment) | within 2 weeks of patient completion of treatment
  Patient completion of questionnaire to determine acceptance and tolerability of immobilisation shell during fabrication (moulding) and planning CT scan. All three patient questionnaires will be analysed separately and together to determine any differences between both groups.
Patient acceptance and tolerability of immobilisation shells (1st fraction) | within 2 weeks of patient completion of treatment
  Patient completion of questionnaire to determine acceptance and tolerability of immobilisation shell during first radiotherapy treatment session. All three patient questionnaires will be analysed separately and together to determine any differences between both groups.
Patient acceptance and tolerability of immobilisation shells (last fraction) | within 2 weeks of patient completion of treatment
  Patient completion of questionnaire to determine acceptance and tolerability of immobilisation shell during last radiotherapy treatment session. All three patient questionnaires will be analysed separately and together to determine any differences between both groups.
Radiographer satisfaction of using immobilisation shells (pre-treatment) | within 2 weeks of patient completion of treatment
  Radiographer completion of questionnaire to determine satisfaction with fabrication and use of immobilisation shell during pre-treatment stages. Pre-treatment and treatment questionnaires will be analysed individually and together to determine any differences between both groups.
Radiographer satisfaction of using immobilisation shells (treatment) | within 2 weeks of patient completion of treatment
  Radiographer completion of questionnaire to determine satisfaction with use of immobilisation shell during treatment. The same questionnaire is used at the first and last fraction of treatment. Pre-treatment and treatment questionnaires will be analysed individually and together to determine any differences between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Liam Welsh, PhD, FRCR, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication
Supporting Information: Study Protocol, ICF
Time Frame: Starting 6 months after publication for a period of one year.
Access Criteria: Requests via corresponding author for interested parties working in the field of Radiation Oncology. Information will be shared by corresponding author.